CLINICAL TRIAL: NCT05665699
Title: A Randomized, Open-Label, Multiple-Dose Phase II Study to Evaluate Efficacy and Safety of D-0120 Administered in Combination With Allopurinol in Subjects With Gout
Brief Title: Phase II Study to Evaluate Efficacy and Safety of D-0120 in Combination With Allopurinol in Subjects With Gout
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0120-205
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-08

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Intervention Model Description: Randomized , Open Label, Multiple Dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): week 1: D-0120 low dose in combination with Allopurinol week 2-12: D-0120 increased dose in combination with Allopurinol
  Interventions: Drug: D-0120; Drug: Allopurinol
- Cohort B (Experimental): week 1: D-0120 low dose in combination with Allopurinol week 2: D-0120 increased dose in combination with Allopurinol week 3-12: D-0120 high dose in combination with Allopurinol
  Interventions: Drug: D-0120; Drug: Allopurinol

INTERVENTIONS:
Drug: D-0120 — increasing dose of D-0120
Drug: Allopurinol — standard dosing

SUMMARY:
D-0120 is being tested in combination with Allopurinol in adult subjects with Gout.

ELIGIBILITY:
Inclusion Criteria:

* Gout subjects meeting 2015 ACR/EULAR Gout Classification Criteria with inadequate urate-lowering response
* Subject has had at least 2 gout flares in the previous 12 months.
* Body Mass Index (BMI) between 18.0 and 45.0 kg/m2 (inclusive).
* Male and Female Subjects must agree to abstain or use effective contraception methods from the time of signing ICF and for the duration of study participation through 30 days after the last dose of study drug.
* Subjects must have adequate clinical laboratory and ECG results as assessed by the Principal Investigator

Exclusion Criteria:

* Subjects with significant comorbidities, inadequate lab function, current (and within the past 5 years) diagnosis of cancer or any condition that, in the judgment of the investigator, would place him/her at undue risk, or potentially compromise the results or interpretation of the study.
* Women who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
• To assess the efficacy of D-0120 in combination with allopurinol to reduce serum urate levels in treatment of patients with gout by week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Stazzone, Study Director — InventisBio Co., Ltd
Locations (19):
- United States (19):
  - Study Center, Birmingham, Alabama
  - Site Center, Plantation, Florida
  - Study Center, Evergreen Park, Illinois
  - Study Center, Brownsburg, Indiana
  - Site Center, Louisville, Kentucky
  - Study Center, Hickory, North Carolina
  - Study Center, Rocky Mount, North Carolina
  - Study Center, Salisbury, North Carolina
  - Study Center, Wilmington, North Carolina
  - Study Center, Winston-Salem, North Carolina
  - Study Center, Scottdale, Pennsylvania
  - Study Center, Bristol, Tennessee
  - Site Center, Hendersonville, Tennessee
  - Study Center, Knoxville, Tennessee
  - Site Center, Fort Worth, Texas
  - Site Center, The Woodlands, Texas
  - Site Center, Richmond, Virginia
  - Site Center, Bellevue, Washington
  - Study Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No